CLINICAL TRIAL: NCT01454271
Title: Follow up Study of Patients Undergoing Total Hip Arthroplasty CERAFIT® Grafted With Poly Sodium Styrene Sulfonate
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We have decided to design a comparative study which is ongoing
Sponsor: Societe ACTIVBIOMAT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERAVERBIO11; 2011-A00597-34 (Other: AFSSAPS)
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Hip Arthroplasty Replacement
Keywords: Total Hip arthroplasty; Hip Osteoarthritis; Infection after Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total Hip Arthroplasty CERAFIT® grafted (Experimental)
  Interventions: Procedure: Total Hip Arthroplasty Replacement

INTERVENTIONS:
Procedure: Total Hip Arthroplasty Replacement — Total Hip Arthroplasty Replacement

SUMMARY:
The risk of infection after primary Total Hip Arthroplasties (THA)is generally estimated to be less than 1% but remains a severe and costly complication, source of morbidity and even mortality. The "biofilm" forms very early after the bacterial contamination of the prosthesis and poses a number of clinical challenges due to his resistance to immune defence mechanisms and antibiotics. Preventive strategies are needed. The poly sodium styrene sulfonate (pNaSS) is a bioactive polymer. In vitro and in vivo studies showed that poly sodium styrene sulfonate grafted on titane surfaces reduce significantly the bacterial adhesion. They also proved his biocompatibility and osseous-integration.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 75 years old
* Aetiologies for THA : primary osteoarthritis, inflammatory diseases,Osteonecrosis

Exclusion Criteria:

* Previous infectious hip arthritis
* Previous surgeries on the operated hip
* Revision of THA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Femoral component osseous-integration | 1 year after surgery
  Scoring system of Engh

SECONDARY OUTCOMES:
Infection rate | 1 year after surgery
  Infection (yes/no) :
  Clinical, biological or radiological THA infection signs. In the case of infection suspicion, hip aspiration will be performed with joint fluid culture
Quality of Life | One, three, six and twelve months after surgery
  SF-36 score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Hardy, Ph.D., Principal Investigator — Ambroise Paré Hospital
Locations (1):
- Ambroise Paré Hospital. Orthopaedic surgery department, Boulogne-Billancourt, Île-de-France Region, France